CLINICAL TRIAL: NCT06915623
Title: Nanocrystal Gels to Treat and Prevent Peri-implant Mucositis: A Randomized Controlled Pilot Study
Brief Title: Gels to Treat and Prevent Gingival Inflammation Around Dental Implants
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nancy Mouradian (Other)
Collaborators: Invicare Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Nancy Mouradian, Doctor, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-257 A-3/13-04-2023
Record Dates: First submitted 2025-03-28; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Peri-implant Mucositis; Healthy Peri-implant
Keywords: Peri-implant mucositis; clinical trial; pilot study; healthy peri-implant; bleeding on probing; nanocrystal gel

STUDY DESIGN:
Intervention Model Description: Test group: Received standard intervention and Gel intervention Control group: Received standard intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): This group received standard mechanical debridement around the implants with a nanocrystal gel administered topically as an adjunct treatment.
  Interventions: Drug: Innovative Gel application; Procedure: Mechanical Debridement
- Control group (Active Comparator): This group only received standard mechanical debridement around implants.
  Interventions: Procedure: Mechanical Debridement

INTERVENTIONS:
Drug: Innovative Gel application — Innovative gel application: Gel is applied as an adjunct treatment to cleaning and scaling.
  Arms: Test Group
Procedure: Mechanical Debridement — Cleaning and scaling of the implant.

SUMMARY:
This study aims to evaluate a gel's potential to improve gum health around dental implants when used alongside traditional cleaning methods. The central research question is:

Does the gel reduce gum bleeding?

Researchers will compare the effects of traditional dental cleaning alone wit those of dental cleaning combined with gel administration, focusing on overall gum health around implants. The study will enroll eight participants-some with early gum issues, such as bleeding gums, and others with healthy gums. Each participant will be randomly assigned to receive either regular dental cleaning or the cleaning paired with gel application.

The study process includes the following steps:

1. Participants will visit the clinic and receive one of the two treatments randomly.
2. One week later, they will complete a printed survey detailing any symptoms or discomfort experienced .
3. After four weeks, participants will return to the clinic for checkups and tests to measure progress.

DETAILED DESCRIPTION:
This clinical study, conducted at Laval University's graduate periodontics clinic, investigates the efficacy and safety of a nanocrystal gel as a supplementary treatment to non-surgical mechanical debridement (professional cleaning) for managing peri-implant mucositis-a reversible inflammatory condition affecting the soft tissues around dental implants. The study enrolls eight participants, comprising individuals with either healthy peri-implant tissues or peri-implant mucositis. Participants are randomly assigned to one of two groups: the test group receives the nanocrystal gel in conjunction with standard peri-implant therapy, while the control group undergoes peri-implant therapy alone.

The primary focus of the investigation is the bleeding on probing (BoP) parameter, analyzing its progression over a four-week period and comparing outcomes between the two groups. Additionally, other clinical parameters, including the modified gingival index, modified plaque index, and pocket depth, are evaluated.

Participants receive one of the designated treatments, with the study design ensuring they are blinded to the specific treatment administered. A follow-up appointment four weeks later allows for the reassessment of all recorded clinical parameters. One week after treatment, participants complete a survey to report any discomfort or pain experienced post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Maxillary or mandibular fixed implant-supported prostheses (up to 3 units)
* Diagnosis of peri-implant health or peri-implant mucositis
* Signed an informed consent form

Exclusion Criteria:

* Advanced peri-implantitis
* Extensive implant-supported restorations (four units or more)
* Recent radiotherapy, chemotherapy, long-term systemic corticosteroid therapy
* Drugs inducing gingival hyperplasia
* Recent antibiotics (within three months)
* Prosthetic restorations impeding clinical assessment
* Poor marginal contours or prosthetic complications
* Peri-implant bone loss exceeding 30%
* Acute oral infection
* Uncontrolled diabetes, systemic diseases, immune deficiency, autoimmune disease
* Long-term bisphosphonate use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | First assessment is the day of the intervention and the last one is 4 weeks later at follow-up.
  A periodontal probe is gently inserted into the sulcus (the space between the implant and the surrounding gum tissue). The probe is moved around the implant in a sweeping motion, covering all surfaces (Mesial, Distal, Buccal and Palatal/Lingual). This gesture is done with light pressure to avoid causing unnecessary trauma to the tissues. After probing, the clinician observes the site for any bleeding. Bleeding that occurs within 10 to 15 seconds after probing is recorded as a positive BOP result.

SECONDARY OUTCOMES:
Plaque index (PI) | It is assessed on intervention day and at a 4 week- follow up appointment
  The plaque index is calculated by assigning a score to each surface based on the presence of plaque present, after probing. It is registered on the Mesial, Distal, buccal and palatal/lingual sides of the implant. Scores are reported dichotomously. It categorizes plaque as either present or absent, using a binary scoring system:
  1: Presence of plaque 0: Absence of plaque A higher overall plaque score could indicate a worse outcome with a higher risk of inflammation of the tissues surrounding the implant.
Modified Gingival Index (MGI) | It is assessed on intervention day and at a 4 week- follow up appointment
  The testing was made similarly to the bleeding on probing, but also takes into consideration the visual evaluation of the tissues around the implant. The clinician focuses on detecting visual signs of inflammation, such as redness, swelling, and altered gingival contour. It is tested on the mesial, distal, buccal and palatal/lingual sides of the implant. Results are reported from a 0 to 4 scale with 0 indicating no bleeding and 4 indicating extreme inflammation with ulceration and tissue damage.
Probing Depth | It is assessed on intervention day and at a 4 week- follow up appointment
  It is measured using a UNC15 periodontal probe. It is gently inserted into the sulcus or pocket surrounding the implant, following the contours of the implant and tissue. Care is taken to avoid excessive pressure, which could damage the delicate peri-implant tissue or lead to inaccurate readings. It is assessed at the mesial, distal, buccal and palatal/lingual sides.

OTHER OUTCOMES:
Suppuration | It's assessed at the 4 week follow-up appointment.
  Presence or Absence were noted (qualitatively) 15 seconds after probing test.
Irritation, Pain and Discomfort | This was reported at 7 days post-op.
  These are subjective outcomes reported by the patient by a questionnaire sent to them. Patients have to indicate from a scale of 0 to 10 :
  * Discomfort (0 is no discomfort and 10 is the worst discomfort)
  * Irritation (0 is no irritation and 10 is the worst irritation)
  * Pain (0 is no pain and 10 is the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Mouradian, DMD, MSc, FRCD(C), Dip.ABP, Study Director — Laval University; Beatrice Groleau-Asselin, DMD, MSc, FRCD(C), Principal Investigator — Laval University
Locations (1):
- Faculté de Médecine dentaire de l'Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
In the patient consent form, possible IPD sharing was not disclosed. This might be considered in future trial registrations.

REFERENCES:
- [Background] Tamimi F, Le Nihouannen D, Bassett DC, Ibasco S, Gbureck U, Knowles J, Wright A, Flynn A, Komarova SV, Barralet JE. Biocompatibility of magnesium phosphate minerals and their stability under physiological conditions. Acta Biomater. 2011 Jun;7(6):2678-85. doi: 10.1016/j.actbio.2011.02.007. Epub 2011 Feb 13. PMID 21324383
- [Background] Laurenti M, Al Subaie A, Abdallah MN, Cortes AR, Ackerman JL, Vali H, Basu K, Zhang YL, Murshed M, Strandman S, Zhu J, Makhoul N, Barralet JE, Tamimi F. Two-Dimensional Magnesium Phosphate Nanosheets Form Highly Thixotropic Gels That Up-Regulate Bone Formation. Nano Lett. 2016 Aug 10;16(8):4779-87. doi: 10.1021/acs.nanolett.6b00636. Epub 2016 Jul 6. PMID 27280476
- [Background] Figuero E, Graziani F, Sanz I, Herrera D, Sanz M. Management of peri-implant mucositis and peri-implantitis. Periodontol 2000. 2014 Oct;66(1):255-73. doi: 10.1111/prd.12049. PMID 25123773
- [Background] Behmanesh S, Chow K, Dondani J, Al-Hashedi A, Tamimi F. Effectiveness of 2D magnesium phosphate hydrogel for surgical decontamination of dental implants: A case series. J Prosthodont. 2025 Jun;34(5):449-455. doi: 10.1111/jopr.13961. Epub 2024 Oct 3. PMID 39363547
- [Background] Al-Hashedi AA, Laurenti M, Benhamou V, Tamimi F. Decontamination of titanium implants using physical methods. Clin Oral Implants Res. 2017 Aug;28(8):1013-1021. doi: 10.1111/clr.12914. Epub 2016 Jul 8. PMID 27392811